CLINICAL TRIAL: NCT03113500
Title: A Phase 2 Study of Brentuximab Vedotin Plus Cyclophosphamide, Doxorubicin, Etoposide, and Prednisone (CHEP-BV) Followed by BV Consolidation in Patients With CD30-Positive Peripheral T-Cell Lymphomas
Brief Title: Brentuximab Vedotin and Combination Chemotherapy in Treating Patients With CD30-Positive Peripheral T-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17058; NCI-2017-00573 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17058 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Adult T-Cell Leukemia/Lymphoma; Anaplastic Large Cell Lymphoma, ALK-Negative; Anaplastic Large Cell Lymphoma, ALK-Positive; Angioimmunoblastic T-Cell Lymphoma; Ann Arbor Stage II Noncutaneous Anaplastic Large Cell Lymphoma; Ann Arbor Stage III Noncutaneous Anaplastic Large Cell Lymphoma; Ann Arbor Stage IV Noncutaneous Anaplastic Large Cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Hepatosplenic T-Cell Lymphoma; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, T-Cell | interventions — Brentuximab Vedotin; Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CHEP-BV) (Experimental): INDUCTION: Patients receive cyclophosphamide IV and doxorubicin IV on day 1, etoposide IV on days 1-3, and prednisone PO on days 1-5. Patients also receive brentuximab vedotin IV over approximately 30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (or for up to 5 cycles for patients who received 1 cycle of CHOP-like or CHP-BV therapy prior to induction, per investigator's discretion) in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Between 30-60 days post-consolidative autologous stem cell therapy, post-consolidative radiation therapy, or after completing induction cycle 6 (cycle 5 for patients who qualify for receiving 5 cycles of CHEP-BV instead of 6), patients with objective response (complete response or partial response) receive brentuximab vedotin IV over approximately 30 minutes on day 1. Treatment repeats every 21 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Etoposide Phosphate; Other: Laboratory Biomarker Analysis; Drug: Prednisone

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone

SUMMARY:
This phase II trial studies the side effects and how well brentuximab vedotin and combination chemotherapy work in treating patients with CD30-positive peripheral T-cell lymphoma. Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in a targeted way and delivers vedotin to kill them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, etoposide, and prednisone work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving brentuximab vedotin and combination chemotherapy may work better in treating patients with CD30-positive peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of cyclophosphamide, doxorubicin hydrochloride (doxorubicin), etoposide phosphate (etoposide), prednisone, and brentuximab vedotin (CHEP-BV), as induction therapy in patients with CD30-positive peripheral T-cell lymphoma (PTCL). (Safety lead-in) II. Assess the anti-lymphoma activity of CHEP-BV as induction treatment in patients with CD30-positive PTCL. (Phase 2)

SECONDARY OBJECTIVES:

I. Describe outcomes of CD30-positive PTCL patients who go on to receive BV consolidation therapy post CHEP-BV induction with/without autologous hematopoietic cell transplantation/radiation.

EXPLORATORY OBJECTIVES:

I. Explore the rate of minimal residual disease (MRD) negativity (as assessed by next-generation sequencing) and MRD kinetics after CHEP-BV and BV consolidation therapy in CD30-positive PTCL.

II. Explore the possible association between outcome after study treatment and CD30 expression, gene expression profiles (GEP), and genetic mutations as measured in PTCL tumor samples.

OUTLINE:

INDUCTION: Patients receive cyclophosphamide intravenously (IV) and doxorubicin IV on day 1, etoposide IV on days 1-3, and prednisone orally (PO) on days 1-5. Patients also receive brentuximab vedotin IV over approximately 30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (or for up to 5 cycles for patients who received 1 cycle of cyclophosphamide, doxorubicin, vincristine and prednisone [CHOP]-like or brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone [CHP-BV] therapy prior to induction, per investigator's discretion) in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Between 30-60 days post-consolidative autologous stem cell therapy, post-consolidative radiation therapy, or after completing induction cycle 6 (cycle 5 for patients who qualify for receiving 5 cycles of CHEP-BV instead of 6), patients with objective response (complete response or partial response) receive brentuximab vedotin IV over approximately 30 minutes on day 1. Treatment repeats every 21 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of participant and/or legally authorized representative
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies will be retrieved and submitted post-enrollment

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* Eastern Cooperative Oncology Group (ECOG) status =< 2
* Histologically confirmed mature peripheral T-cell or natural killer (NK)-cell lymphoma per World Health Organization (WHO) classification, including:

  * Anaplastic lymphoma kinase (ALK)-positive anaplastic large cell lymphoma (ALCL) with international protein index (IPI) of 2 or higher (must have bulky [defined as mass >= 10 cm] stage II, or stage III-IV disease)
  * ALK-negative ALCL

    * NOTE: Per amendment dated 05-10-19, ALCL will no longer be eligible except for Canada.
  * PTCL-not otherwise specified (NOS)
  * Angioimmunoblastic T-cell lymphoma (AITL)
  * Adult T-cell lymphoma/leukemia (ATLL)
  * Enteropathy-associated T-cell lymphoma (EATL)
  * Hepatosplenic T-cell lymphoma
* CD30-positivity (e.g. at least 1%) by immunohistochemistry confirmed by hematopathology review at the participating institution
* Measurable disease of at least 1.5 cm on computed tomography (CT) or positron emission tomography (PET)-CT scan
* Absolute neutrophil count (ANC) >= 1,000/mm^3

  * Exception: unless documented bone marrow involvement by lymphoma
* Platelets >= 50,000/mm^3

  * Exception: unless documented bone marrow involvement by lymphoma
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN) OR if hepatic involvement by lymphoma: =< 3 x ULN for Gilbert's disease or documented hepatic involvement by lymphoma
* Aspartate aminotransferase (AST) =< 2 x ULN OR if hepatic involvement by lymphoma: AST =< 5 x ULN
* Alanine aminotransferase (ALT) =< 2 x ULN OR if hepatic involvement by lymphoma: ALT =< 5 x ULN
* Creatinine clearance of >= 60 mL/min per the Cockcroft-Gault formula
* Left ventricular ejection fraction (LVEF) >= 45%
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by WOCBP and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy; childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior treatment of PTCL with systemic anti-lymphoma therapies, investigational agents, radiation

  * Exception: May have received 1 cycle of CHOP-like therapy (e.g. CHOP, CHOEP, EPOCH) or 1 cycle of CHP-BV; these participants must initiate day 1 cycle 1 of study therapy (CHEP-BV) no less than 19 days from prior CHOP-like or CHP-BV therapy; Patients who received 1 cycle of CHOP-like or 1 cycle of CHP-BV therapy prior to initiating induction with CHEP-BV are allowed to receive only 5 cycles of CHEP-BV instead of 6 cycles, per investigator's discretion
* History of another primary invasive cancer, hematologic malignancy, or myelodysplastic syndrome that has not been in remission for at least 3 years.

  * Exceptions: Non-melanoma skin cancer and in situ cervical cancer
* Symptomatic cardiac disease (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias), cerebrovascular event/stroke or myocardial infarction within the past 6 months
* Central nervous system involvement by lymphoma, including leptomeningeal involvement
* History of progressive multifocal leukoencephalopathy (PML)
* Active >= grade 3 viral, bacterial, or fungal infection within 2 weeks prior to day 1 of protocol therapy
* Any known human immunodeficiency virus (HIV) infection, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Baseline peripheral neuropathy >= grade 2 or patients with the demyelinating form of Charcot-Marie-Tooth syndrome
* Known severe hypersensitivity to any study related agent excipient(s)
* Females only: pregnant or breastfeeding
* Any other condition that would, in the investigator's judgement, contraindicate the patient's participation in the clinical study
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2026-07-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (5):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas
- BCCA-Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Herrera AF, Zain J, Savage KJ, Feldman T, Brammer JE, Chen L, Puverel S, Popplewell L, Budde LE, Mei M, Hosing C, Nair R, Leslie L, Daniels S, Peters L, Forman S, Rosen S, Kwak L, Iyer SP. Brentuximab vedotin plus cyclophosphamide, doxorubicin, etoposide, and prednisone followed by brentuximab vedotin consolidation in CD30-positive peripheral T-cell lymphomas: a multicentre, single-arm, phase 2 study. Lancet Haematol. 2024 Sep;11(9):e671-e681. doi: 10.1016/S2352-3026(24)00171-6. Epub 2024 Jul 24. PMID 39067464

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (CHEP-BV): INDUCTION: Patients receive cyclophosphamide IV and doxorubicin IV on day 1, etoposide IV on days 1-3, and prednisone PO on days 1-5. Patients also receive brentuximab vedotin IV over approximately 30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (or for up to 5 cycles for patients who received 1 cycle of CHOP-like or CHP-BV therapy prior to induction, per investigator's discretion) in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Between 30-60 days post-consolidative autologous stem cell therapy, post-consolidative radiation therapy, or after completing induction cycle 6 (cycle 5 for patients who qualify for receiving 5 cycles of CHEP-BV instead of 6), patients with objective response (complete response or partial response) receive brentuximab vedotin IV over approximately 30 minutes on day 1. Treatment repeats every 21 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Brentuximab Vedotin: Given IV
  Cyclophosphamide: Given IV
  Doxorubicin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Etoposide Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Prednisone: Given PO
Period: Overall Study
Arm/Group | Treatment (CHEP-BV)
Started | 48
Completed | 47
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (CHEP-BV)
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 56 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate After Cyclophosphamide, Doxorubicin, Etoposide, Prednisone, and Brentuximab Vedotin (CHEP-BV) Induction Therapy
Description: CR rate was estimated by the proportion of evaluable patients achieving CR after CHEP-BV induction therapy, along with the 95% exact binomial confidence interval.
Time Frame: Up to the end of the CHEP-BV treatment
Population: 1 subject had no disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of response rate
Arm/Group | Treatment (CHEP-BV)
Number analyzed (Participants) | 47
percentage of response rate | 79 [64 to 89]

2. Secondary Outcome: Overall Survival at 1 Year
Description: Overall survival (OS) was measured from enrollment to death from any cause. OS was estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error.
Time Frame: The time from enrollment to death from any cause assessed up to 1 year.
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Treatment (CHEP-BV)
Number analyzed (Participants) | 48
percentage of survival probability | 91 [78 to 97]

ADVERSE EVENTS:
Time Frame: Up to 30 days post treatment
Arm/Group | Treatment (CHEP-BV)
All-Cause Mortality (participants affected / at risk) | 1/48
Serious Adverse Events (participants affected / at risk) | 22/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (CHEP-BV) (N=48)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (13)
eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
perforated sigmoid diverticulitis (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 6 (9)
Infection, NOS (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
c. septicum infection (Infections and infestations) | 1 (1)
c.diff infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (CHEP-BV) (N=48)
Anemia (Blood and lymphatic system disorders) | 33 (148)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (11)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (3)
Palpitations (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 5 (8)
Sinus tachycardia (Cardiac disorders) | 13 (30)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (2)
ear wax (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 6 (8)
Conjunctivitis (Eye disorders) | 3 (3)
Dry eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 2 (2)
Itching Around Eyes (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 3 (3)
blepharitis (Eye disorders) | 1 (1)
eye fatigue (Eye disorders) | 1 (1)
puffy eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 15 (22)
Anal ulcer (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Blood In Stools (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 17 (40)
Diarrhea (Gastrointestinal disorders) | 19 (32)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Hemorrhoids (Gastrointestinal disorders) | 4 (5)
Mucositis oral (Gastrointestinal disorders) | 17 (29)
Nausea (Gastrointestinal disorders) | 34 (87)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (25)
blood in stool (Gastrointestinal disorders) | 1 (1)
tarry stools (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 6 (10)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 39 (105)
Fever (General disorders) | 14 (18)
Flu like symptoms (General disorders) | 3 (3)
Gait disturbance (General disorders) | 6 (7)
Infusion related reaction (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (2)
Malaise (General disorders) | 8 (11)
Non-cardiac chest pain (General disorders) | 4 (4)
Pain (General disorders) | 9 (15)
back paresthesia (General disorders) | 1 (1)
coated tounge (General disorders) | 1 (1)
cold sore (General disorders) | 1 (1)
muscle pain (General disorders) | 1 (1)
spleen paresthesia (General disorders) | 1 (1)
tongue sensitivity (General disorders) | 1 (1)
lymphomatoid papulosis (Immune system disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
DIFF INFECTION (Infections and infestations) | 1 (1)
DIFFICILE (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Other; Bacteremia (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 4 (7)
Strep bacteremia (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 7 (9)
Urinary tract infection (Infections and infestations) | 3 (6)
gram positive cocci infection (Infections and infestations) | 1 (1)
oral thrush (Infections and infestations) | 1 (2)
shingles (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (6)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (15)
Alanine aminotransferase increased (Investigations) | 18 (58)
Alkaline phosphatase increased (Investigations) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 17 (36)
Blood bilirubin increased (Investigations) | 9 (9)
CD4 lymphocytes decreased (Investigations) | 4 (7)
CPK increased (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 6 (22)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Elevated Lactic Acid (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Increased white blood cells (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 23 (80)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 27 (72)
Platelet count decreased (Investigations) | 24 (79)
Serum amylase increased (Investigations) | 2 (2)
Weight gain (Investigations) | 7 (25)
Weight loss (Investigations) | 7 (13)
White blood cell decreased (Investigations) | 21 (59)
Anorexia (Metabolism and nutrition disorders) | 12 (22)
Dehydration (Metabolism and nutrition disorders) | 5 (7)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (18)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (12)
Hypokalemia (Metabolism and nutrition disorders) | 16 (24)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (19)
Hyponatremia (Metabolism and nutrition disorders) | 15 (30)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (18)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 3 (9)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (11)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot drop (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Interscapular pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (29)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 18 (29)
Dysgeusia (Nervous system disorders) | 7 (9)
Headache (Nervous system disorders) | 13 (21)
Memory impairment (Nervous system disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 2 (2)
Parathesia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 5 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (135)
Presyncope (Nervous system disorders) | 1 (2)
Tingling sensation in fingers/feet (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 8 (11)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 6 (7)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 12 (33)
Personality change (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep disturbance (Psychiatric disorders) | 1 (1)
intermittent mood changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Difficulty with urination (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
dysuria (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (26)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Changes (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Abcess (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (18)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (17)
Skin Flare Reaction (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin tear on knuckle (Skin and subcutaneous tissue disorders) | 1 (1)
blood at the surface of skin (Skin and subcutaneous tissue disorders) | 1 (1)
brittle nails (Skin and subcutaneous tissue disorders) | 1 (1)
night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
papular rash on back and arms (Skin and subcutaneous tissue disorders) | 1 (1)
skin injury (Skin and subcutaneous tissue disorders) | 1 (1)
skin lesion on left lateral thigh (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 14 (76)
Hypotension (Vascular disorders) | 10 (16)
Thromboembolic event (Vascular disorders) | 3 (9)
vascular access complication (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT03113500/Prot_SAP_000.pdf